CLINICAL TRIAL: NCT01450891
Title: Novel Diagnostic Approaches for the Diagnosis of Alzheimer's Disease: Technology Assessment and Clinical Effectiveness
Brief Title: Health Technology Assessment of Diagnostic Approaches in Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Center for Translational Molecular Medicine (Other); Leiden University Medical Center (Other); Radboud University Medical Center (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: Sponsor
Other Study IDs: 09-3-038; 02N-101 (Other Grant/Funding Number: Center for Translational Molecular Medicine (CTMM))
Record Dates: First submitted 2011-09-20; First posted 2011-10-12 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Neurodegenerative Diseases; Memory Disturbances
Keywords: Alzheimer's disease; Diagnosis; Costs; Benefits; subjective and/or objective memory complaints
MeSH Terms: conditions — Neurodegenerative Diseases; Alzheimer Disease; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cerebrospinal fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- total patient group: all new consecutive patients of the participating memory clinics who are suspected of having a primary neurodegenerative disease, meaning that all patients with subjective as well as objective memory complaints are included

SUMMARY:
Background: New research criteria for the diagnosis of Alzheimer's disease (AD) have recently been developed to enable an early diagnosis of AD pathophysiology by relying on emerging biomarkers. To enable efficient allocation of health care resources, evidence is needed to support decision makers on the adoption of emerging biomarkers in clinical practice. The research goals are to 1) assess the diagnostic test accuracy (of current clinical diagnostic work-up and emerging biomarkers in Magnetic Resonance Imaging (MRI), Positron Emission Tomography (PET) and Cerebrospinal Fluid (CSF), 2) perform a cost-consequence analysis and 3) assess long-term cost-effectiveness by an economic model.

Methods/design: In a cohort design 304 consecutive patients suspected of having a primary neurodegenerative disease are approached in four academic memory clinics and followed for two years. Clinical data and data on quality of life data, costs and emerging biomarkers are gathered.

Diagnostic test accuracy is determined by relating the clinical practice and new research criteria diagnoses to the reference diagnosis. The clinical practice diagnosis at baseline is reflected by a consensus procedure among experts using clinical information only (no biomarkers). The diagnosis based on the new research criteria is reflected by decision rules that combine clinical and biomarker information. The reference diagnosis is determined by a consensus procedure among experts based on clinical information on the course of symptoms over a two-year time period.

A decision analytic model is build combining available evidence from different resources among which (accuracy) results from the study, literature and expert opinion to assess long-term cost-effectiveness of the emerging biomarkers.

Discussion: Several other multi-centre trials study the relative value of new biomarkers for early evaluation of AD and related disorders. The uniqueness of this study is the assessment of resource utilization and quality of life to enable an economic evaluation. The study results are generalizable to a population of patients who are referred to a memory clinic due to their memory problems.

ELIGIBILITY:
Inclusion Criteria:

* All new consecutive patients of the participating memory clinics who are suspected of having a primary neurodegenerative disease. This means all patients with subjective and/or objective memory complaints.
* CDR 0, 0.5 or 1
* MMSE score must be 20 or higher.
* Availability of a reliable informer or proxy (who visits or contacts the patient at least once a week).

Exclusion Criteria:

* Normal Pressure Hydrocephalus (NPH)
* Huntington's disease
* Recent Transient Ischaemic Attack (TIA) (<2 years) or Cerebral Vascular Accident (CVA) or TIA/CVA followed by cognitive impairment (within 3 months)
* History of Schizophrenia, other psychotic disorders (< 12 months)
* Major depression (< 12 months)
* Alcohol abuse
* Brain-tumor, epilepsy, encephalitis
* Absence of a reliable informant
* Probably not available for follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 304 consecutive patients, of four academic memory clinics specialized in the diagnosis and treatment of memory disorders, who were suspected of having a primary neurodegenerative disease were approached for participating in the study. This included all patients with subjective and/or objective memory complaints. Eligibility criteria were chosen to represent current clinical situation and enable generalisability to clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2009-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of Magnetic Resonance Imaging (MRI) | baseline
  Diagnostic test accuracy (in terms of sensitivity and specificity) of three MRI markers (Whole brain and hippocampal volume, white matter integrity, and functional connectivity) is determined by relating the particular marker to a reference diagnosis. The reference diagnosis is determined by a consensus procedure among experts based on clinical information on the course of symptoms over a two-year time period.
Change in cognition at 2 years | baseline, 1 year follow up, 2 year follow up
  Measured by the Mini-mental state examination (MMSE).
Change in dementia severity at 2 years | baseline, 1 year follow up, 2 year follow up
  Measured by the clinical dementia rating (CDR) scale.
Change in quality of life at 2 years | baseline, 3 months follow up, 1 year follow up, 2 year follow up
  Measured by the Euro-Qol-5D both by the patient and caregiver and measured by the Quality of life Alzheimer's disease state (QoL-AD) both by the patient and caregiver.
Health care resource use during 2 years | baseline, 3 months follow up, 1 year follow up, 2 year follow up
  By means of questionnaires the health care resource usage is measured by the Resource Utilization in Dementia-questionnaire (RUD-lite) over a period of 2 years using 4 measurement moments to interpolate the data.
Change in productivity at 2 years | baseline, 3 months follow up, 1 year follow up, 2 year follow up
  Work status, income, and productivity losses of both the patient and caregiver are assessed by the adjusted PRODISQ (PROductivity and DISease Questionnaire). The consequences of informal caregiving on paid or unpaid work are assessed by the Health and Labour Questionnaire.
Diagnostic accuracy of cerebrospinal fluid (CSF) | baseline
  Diagnostic test accuracy (in terms of sensitivity and specificity) of three CSF markers (CSF total tau, CSF phosphorylated tau, and CSF Aβ1-42) is determined by relating the particular marker to a reference diagnosis. The reference diagnosis is determined by a consensus procedure among experts based on clinical information on the course of symptoms over a two-year time period.

SECONDARY OUTCOMES:
Demographic changes at 2 years | baseline, 1 year follow up, 2 year follow up
  Course of cognitive symptoms, Civil status, and Living situation are assessed.
General clinical changes at 2 years | baseline, 1 year follow up, 2 year follow up
  Smoking behaviour, alcohol intake, length, weight, blood pressure, neuropsychological problems, and co-morbidities are assessed.
Change in behavioural and psychological problems at 2 years | baseline, 1 year follow up, 2 year follow up
  Measured by the Neuropsychiatric Inventory (NPI).
Change in basic and instrumental activities in daily activities at 2 years | baseline, 1 year follow up, 2 year follow up
  Measured by the Disability assessment for Dementia (DAD).
Change in depression at 2 years | baseline, 1 year follow up, 2 year follow up
  Measured by the geriatric depression scale 15 (GDS-15).
Change in cognitive functioning at 2 years | baseline, 1 year follow up, 2 year follow up
  A neuropsychological examination is performed using the:
  * Rey's Verbal Learning Test, Visual Association Test, and Digit-Span to assess memory;
  * Letter Digit Substitution Test to assess mental processing rate; and
  * Stroop Color-Word Test and Trail Making Test to assess attention, concentration and interference.
Change in sense of competence at 2 years | baseline, 1 year follow up, 2 year follow up
  Measured by the Sense of Competence Questionnaire (SoCQ).
Change in Care-related quality of life | baseline, 3 months follow up, 1 year follow up, 2 year follow up
  Assessed by the CarerQol by the informal caregiver.

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - VU University Medical Center, Amsterdam
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Center, Maastricht
  - Radboud University Nijmegen Medical Centre, Nijmegen

REFERENCES:
- [Background] Handels RL, Aalten P, Wolfs CA, OldeRikkert M, Scheltens P, Visser PJ, Joore MA, Severens JL, Verhey FR. Diagnostic and economic evaluation of new biomarkers for Alzheimer's disease: the research protocol of a prospective cohort study. BMC Neurol. 2012 Aug 10;12:72. doi: 10.1186/1471-2377-12-72. PMID 22883691
- See also: organizational framework for the study — http://www.ctmm.nl